CLINICAL TRIAL: NCT01304004
Title: Effect of a Drinkable Yogurt Enriched in Proteins and Fibers on Satiety
Acronym: JIVAGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Aliments ULTIMA Foods Inc. (Industry)
Responsible Party: Principal Investigator, Benoit Lamarche, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INAF-2010-154
Record Dates: First submitted 2011-02-22; First posted 2011-02-25 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Obesity
Keywords: Obesity; Yogurt; Proteins; Fibres; Women; Satiety
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental drinking yogurt (Experimental)
  Interventions: Other: Satiety
- Placebo drinking yogurt (Placebo Comparator)
  Interventions: Other: Satiety

INTERVENTIONS:
Other: Satiety — Intervention Description: Consumption of the 2 drinkable yogurts separated by 4 weeks:
  1. Experimental drinkable yogurt enriched in proteins and fibres
  2. Placebo drinkable yogurt (isocaloric and isovolumetric)

SUMMARY:
Worldwide, obesity rate has increased so much in the latest years, that we call it obesity epidemic. Overweight could result of an unbalanced energetic balance for years. The person who regularly consumes more calories than she expends will find herself with a positive energetic balance, which results in a weight gain. A daily overconsumption of only 10 calories comes with a weight gain throughout one year. A way to avoid this overconsumption is to eat food that increases satiety. Satiety can be defined as the time interval after food ingestion, during which hunger and desire to eat are suppressed.

The general objective of the study is to investigate in a pilot study the impact of a drinkable yogurt enriched in proteins and fibres on satiety.

DETAILED DESCRIPTION:
The study will be conducted according to an estimate crossover randomized double-blind and include two treatments to drink that will be tested in each one month apart.

1. Experimental drinkable yogurt enriched in proteins and fibres
2. Placebo drinkable yogurt (isocaloric and isovolumetric)

One the eve of the two tests, participants will consume the same meal at dinner time. During the test days, participants should arrive between 6:30 and 8:30 and will be isolated in a private room suitable for this type of testing. Any reference to time of the day will be eliminated until the end of tests. First, participants will consume a standardized breakfast which corresponds to about 10 to 15% of energy needs of the day. The food provided at breakfast (toast, butter, peanut butter, cheese, orange juice) will be the same in both tests. Participants must consume all food within a period of 15 minutes. Two hours after the start of the test, participants will receive a snack in the form of yogurt (experimental, placebo) they will consume within a period of 5 minutes. Two hours later, participants will receive a lunch buffet consists of food ready to eat. The foods present in the buffet will have an overall energy value of about 1500 kcal, which exceeds the energy needs of participants for this meal. They will be encouraged to consume foods until satiety over a maximum of 30 minutes.

Satiety will be measured by visual analogue scale throughout the test, either immediately before breakfast and snack as well as predetermined times thereafter until the lunch. Participants will have access to water throughout the test. The weight of food consumed and the water intake will be calculated in the absence of the participants and will be used to calculate the energy intake at lunch.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged between 25 and 45 years old
* Body mass index between 20 and 30 kg/m2
* Stable body weight (+/- 2 kg) for 6 months before the beginning of the study
* Smoking or not

Exclusion Criteria:

* Previous history of cardiovascular disease, type 2 diabetes and other endocrine disorders
* High blood pressure (≥ 140/90)
* Previous history of repeated weight loss and weight gain
* Important weight loss during the 6 months before the beginning of the study
* Subjects with high restriction level according to established criteria of a questionnaire that measures restriction level
* Use of natural products or supplements having effects on dietary intake during the 3 months
* Pregnant women
* Subjects taking medications for hypertension, depression, hyperlipidemia or immunosuppressant
* Allergy or intolerance to dairy products
* Vegetarism

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in satiety | Mesured by analogue visual scales at each 30 minutes during 4 hours (for the 2 satiety tests, separeted by four weeks)
  Satiety will be measured by visual analogue scales throughout the test, either immediately before breakfast and snack as well as predetermined times thereafter until the lunch.

SECONDARY OUTCOMES:
Change in energy intake at lunch | Mesured 2 times (during the 2 satiety tests, separeted by four weeks)
  The weight of food consumed and the water intake during the two satiety tests will be calculated in the absence of the participants and will be used to calculate the energy intake at lunch.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît LAmarche, PhD, Principal Investigator — Institute of Nutraceutical and Functional Foods (INAF), Laval University
Locations (1):
- Institute of Nutraceutical and Functional Foods (INAF), Laval University, Québec, Quebec, Canada